CLINICAL TRIAL: NCT06408558
Title: he Effect of Altitude and Simulated Flight in a Hypobaric Chamber on Glucose Metabolism and the in Vivo Performance of Insulin Delivery Systems
Brief Title: Safe Use of New Technologies in Diabetes in Flight
Acronym: SUNDIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Medical University of Graz (Other); KU Leuven (Other); UK Civil Aviation Authority (Unknown); QintetiQ Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FHMS 2022 15
Record Dates: First submitted 2024-04-24; First posted 2024-05-10 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-09

CONDITIONS: Type1 Diabetes
Keywords: Postprandial glucose metabolism
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Intervention Model Description: The study is a randomised crossover study at two different ambient pressures one at normal ambient pressure (760 mmHg) and the other at 560 mmHg mimicking the repressurised cabin environment at 8000 feet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Starting Hypobaric (Experimental): Hypobaric to Ground level & Ground level to Hypobaric
  Interventions: Other: Hypobaric; Other: Ground level
- Starting Ground level (Experimental): Ground level to Hypobaric & Hypobaric to Ground level
  Interventions: Other: Hypobaric; Other: Ground level

INTERVENTIONS:
Other: Hypobaric — The effects of ambient pressure changes on glucose metabolism will be studied
  Other Names: Ambient pressure 560 mmHg
Other: Ground level — The effects of ambient pressure changes on glucose metabolism will be studied
  Other Names: Ambient pressure 760 mmHg

SUMMARY:
Atmospheric pressure can influence how the body handles blood glucose. At high elevations, atmospheric pressure decreases. Research shows that both the elevation and the length of stay at that elevation can influence the body's glucose response.

The investigators would like to find out if the change in pressure in the cabin environment during a flight affects the body's handling of glucose. Commercial planes usually fly at 40000 feet (12192 m) but the cabin pressure is re-pressurized to 8000 feet (2438 m) with cabin pressure fixed at 560 mmHg. The normal atmospheric pressure at sea level is 760 mmHg.

Since the investigators cannot perform the studies in an aeroplane, a hypobaric chamber will be used to set to this low pressure which will reproduce the cabin environment during a commercial flight. The chamber is located at the research and development company, QinetiQ, MOD Boscombe.

The objective of this study is to compare the effect of atmospheric pressure on glucose metabolism during simulated flight conditions during fasting and in response to a mixed liquid meal.

This will involve attending three visits; visit 1 (screening), visit 2 and visit 4 and two phone visits. The duration of the study is 15 days or 1 month depending on the participant's availability. Visit 1, informed consent and screening, will take place at CEDAR, Royal Surrey County Hospital, Guildford, followed by two visits of the meal test in random order at CEDAR or QintetiQ, Visit 2, will be a meal test performed at 760 mmHg OR at 560mmHg. Visit 4, will be a further meal test at 560 mmHg OR 760 mmHg. The order of the meal test visits at different ambient pressures will be randomised. The two phone visits will take place the day after the meal test days to enquire about the patient's health after the test.

DETAILED DESCRIPTION:
The study is a randomised crossover study at two different ambient pressures one at normal ambient pressure (760 mmHg) and the other at 560 mmHg mimicking the repressurised cabin environment at 8000 feet. Participants will have three visits and two phone visits. Visit 1 is the screening visit, Visit 2, will be a meal test (MT) performed at 760 mmHg OR at 560mmHg. Visit 4, will be a further MT at 560 mmHg OR 760 mmHg. The order of MT test visits at different ambient pressures will be randomised. The two phone visits will take place the day after the MT assessment days (visit 3 and 5) with prior arrangement to enquire about the patient's health after the test. The expected duration of participant participation is approximately 15 days.

Screening visit 1 can also be performed before the first test meal on the visit 2 before any visit 2 activities can take place.

Randomisation procedure: The participant will be assigned a study identification number and randomised for the study procedures in random order at different ambient pressures at 760 mmHg and 560 mmHg. Randomisation for the order of the two meal studies, ie at 760 mmHg and at 560mmHg will take place at recruitment phase to accommodate the availability of the volunteers and the dates available at QinetiQ facility for the meal studies.

The recruitment phase will commence as soon as there is ethical, HRA, research governance and regulatory approval and only after the Sponsor 'green light' has been issued.

Recruitment:

* Diabetes Clinics at Cedar centre, Royal Surrey County Hospital.
* And UK CAA Clinic, Aviation House, Gatwick airport.

Identification:

Diabetes Consultants, from diabetes clinics at the CEDAR Centre, Royal Surrey County Hospital will identify participants with type 1 diabetes who are on pump therapy.

The PI will identify participants with type 1 diabetes who are on pump therapy at UK CAA clinic, Gatwick airport at the patient's usual clinic visit.

Screening/run-in period Pilots with type 1 diabetes who are on pump therapy will be approached / recruited at their usual UK-CAA clinic, Aviation House, Gatwick airport by Prof Russell-Jones. Potential participants will be provided with a patient information sheet to take away and read.

Patients with type 1 diabetes who are on pump therapy will be approached and recruited from CEDAR Centre, RSCH. Potential participants will be provided with a patient information sheet to take away and read.

Visit 1: Screening and randomisation (duration 1 h) preformed at visit 1 or upon arrival on the morning of visit The screening and randomisation will take place at CEDAR, RSCH. CEDAR setting: Patients recruited from CEDAR and UK CAA will be invited to a screening visit at CEDAR, RSCH.

Before screening takes place, participants will be provided with verbal and written information about the trial and the procedures involved. The participants will be fully informed of their responsibilities and rights while participating in this trial.

Participants who wish to participate in the trial will be required to sign and date an Informed Consent Form prior to any trial-related activities taking place. The PI on the site will seek informed consent from the participants. All participants will be provided with a copy of the Participant Information Sheet and of their own signed and dated Informed Consent Form.

Demographics: age and sex.

Medical History:

Details of any medical condition or previous condition requiring surgical treatment will be recorded. Including specific questions related to exclusion criteria.

Concomitant Medication

Electrocardiogram (ECG) trace

Physical Examination- Vital Signs Weight (kg), height (cm) and % total body fat mass will be recorded at screening visit and weight only at visit 2 and visit 4. Fat mass using Tanita body composition analyser will only be recorded once at the visit (V2 or V4) taking place at CEDAR using bioimpedance scale Tanita.

Body Mass Index (BMI)

Physical examination will include examination of:

Safety required for hypobaric chamber conditions from QinetiQ will be examined.

Laboratory Tests- plasma HbA1C Randomisation of participant once the eligibility for recruitment to the study is confirmed.

The Metabolic Study- MEAL Test (MT) visit 2 & 4 performed in random order

Participants should refrain from alcohol for 24hours and strenuous exercise for 24 hours prior to any MT assessment day.

The day before the MT. As all participants will be using insulin pump therapy there will be no requirements for any insulin adjustments. The participants will be asked not to consume food and drink only clear fluids from 22.00 the day before the MT until the end of the MT. The participants will attend the clinical research unit, CEDAR, RSCH at Surrey or QinetiQ, MOD Boscombe Down, Wiltshire at 7.00 am the morning of the MT.

The morning of MT- Participants will arrive at QinetiQ or at Cedar centre, at 7 am having fasted overnight. Fasting blood glucose ideally should be between 4 and 8 mmol/L. During the study, the participants' capillary glucose concentration will be measured using a FreeStyle precision Pro, Abbott glucose analyser. The capillary glucose measurements will be recorded against the reading of the CGM glucose monitor. The volume of insulin in the insulin pump will be checked and confirmed at 3ml.

An ECG trace will be performed on the hypobaric visit day (Visit 2 or Visit 4). Blood pressure will be measured at visit 2 and 4.

An intravenous cannula will be inserted in an antecubital fossa of each arm, one for blood sampling and the other for the infusion of the tracer 6,6 2H2 glucose. The blood sampling cannula will be kept patent by flushing with saline after each blood sample (Figure 2). Participants will be asked to empty bladder at -160 min before the study has begun.

At -150 min, baseline blood samples will be taken to measure blood glucose concentration and glucose enrichment by GCMS. Baseline plasma metabolites and hormones will also be measured. Plasma insulin aspart will be measured using an in-house kit at Celerion, Denmark. Glucagon concentration will be measured using radioimmunoassay. Adrenaline and noradrenaline cortisol concentrations will be measured using enzyme linked immunoassays (ELISA).

Having taken the baseline sample, a primed iv infusion of 6, 6 2H2 glucose (6 mg/kg; 0.06mg/kg/min) will commence at -150 min. Blood samples will be taken at 10 min intervals between, -50 min and -30 min and 5 min intervals between -10 min and 0 min. Ambient pressure will start changing at -30 min, reaching decompression pressure at 560 mmHg at -10 min which will remain constant up to 180 min at which time the pressure will be increased gradually to normal pressure at 200min. At 0 min a standardized liquid mixed meal (Ensure; Abbott Nutrition Ohio; 78g carbohydrate consumed within 5 minutes) containing [U-13C] glucose (1.70 g) will be given to measure the meal-derived glucose appearance (11). The participants will be asked to give a standard-wave bolus of insulin where all bolus is delivered at once (0.1U/kg, calculated by investigators) 0-2 minutes before the standard meal test at 0 min. The rate of 6, 6 2H2 glucose infusion will be adjusted at predetermined intervals to mimic the expected endogenous glucose production. Blood sampling will be continued following the meal intake, at regular time points, 10, 20, 30, 60, 75, 90, 120, 150, 180 and 210 min. Infusion of 6, 6 2H2 glucose will be stopped at 180 min.

Vital signs and blood saturation will be measured every 1 h during the MT. Ongoing, the excreted urine volume and glucose concentration in urine will be measured. Urine samples will be analysed for glucose excretion (sugar in the urine) and volume of urine excreted at 0 min before the meal drink and at the end of the study 180 minutes. The urine will be collected at any other time during the study -150 min to 210 min if the patient required to use the toilet. A sample of urine (1 ml) will be centrifuged and stored at -80oC until analysis at a later date at the University of Surrey.

While in the hypobaric chamber blood samples will be kept on ice until centrifugation (Heraeus Labofuge 400 centrifuge, Thermo Fisher Scientific. UK) every 60 min. At CEDAR centre, the MT will be carried out as in the hypobaric chamber but at normal ambient pressure (760 mmHg).

All blood samples will be separated immediately after centrifugation every 60 min and the plasma stored at -20°C at the CEDAR centre overnight and then transferred to a -80°C freezer at the University of Surrey for analysis at a later date at the University of Surrey. The samples from the QinetiQ study day will be stored on dry ice and then transferred to a -80°C freezer at the University of Surrey for analysis at a later date at the University of Surrey.

On completion of the metabolic assessment day, participants will be reminded that they have the telephone number for the research team that can be used 24hours a day.

Atmospheric pressure adjustments In the hypobaric chamber, decompression will start at -30 min and will reach the required 560 mmHg mimicking cabin altitude of 8000 feet in 20 min. The pressure in the chamber will start to increase gradually to 760 mmHg between 180 min and at 200 min a further sample will be taken at the end of study at 210 min.

ELIGIBILITY:
Inclusion Criteria:

* Able in the opinion of the investigator, and willing to give informed consent obtained before any study-related activities.
* Type 1 diabetes
* Duration of type 1 diabetes greater than 12 months.
* Current treatment insulin pump therapy.
* Male or female aged 18 - 65 years.
* BMI of less than 30 kg/m2.
* HbA1c of less than 9%.
* Able and willing to complete the study.
* No cardiovascular complications
* No significant past respiratory disease
* No chronic (long-term) ENT disease such as vertigo, sinusitis or perforated ear drum
* Fitness to undertake long haul airliner flight as a passenger, without assistance or any form of medical support (e.g. supplementary oxygen)
* Patients who are or who have previously been involved in research are eligible provided they have not received an investigational drug within one month of entry into the study

Exclusion Criteria:

* Outside of stated age range.
* Female who is pregnant, breast feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice).
* Participation in any clinical trial of an investigational medicinal product within 30 days before screening.
* Inability to understand verbal and / or written explanations given in English.
* Proliferative retinopathy that has required acute treatment within last three months.
* History of severe renal impairment.
* History of unstable or rapidly progressing renal disease.
* History of hepatic insufficiency / and or significant abnormal liver function.
* Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen and Hepatitis C virus antibody.
* Congestive heart failure defined as New York Heart Association (NYHA) class III and IV, unstable or acute congestive heart failure. Note: eligible patients with congestive heart failure, especially.
* Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Uncontrolled cardiac arrhythmias.
* Uncontrolled hypertension. (BP greater than 160/90).
* Exclude any ENT disease that might interfere with ventilation of the middle ear cavity ('ear clearing') or sinuses
* Any ENT surgery in last 6 months
* Any recent open surgery (last month)
* Claustrophobia
* Inability to communicate over a headset/microphone system
* Intolerance to milk products and those who follow a vegan diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Baseline endogenous glucose production | Through study completion, within 2 years
  Mathematical modelling of the data produced from the isotopic analysis of the samples and glucose concentration (micromol/kg/min)
Postprandial endogenous glucose production | Through study completion, within 2 years
  Mathematical modelling of the data produced from the isotopic analysis of the samples and glucose concentration (micromol/kg/min)
Baseline postprandial glucose uptake | -150 minute to 0 minute during visit 2 and visit 4
  Mathematical modelling of the data produced from the isotopic analysis of the samples and glucose concentration (micromol/kg/min)
Postprandial glucose uptake | Through study completion, within 2 years
  Mathematical modelling of the data produced from the isotopic analysis of the samples and glucose concentration (micromol/kg/min)
Meal derived glucose disposal | Through study completion, within 2 years
  Mathematical modelling of the data produced from the isotopic analysis of the samples and glucose concentration (micromol/kg/min)

SECONDARY OUTCOMES:
Insulin concentration | Through study completion, within 2 years
  Insulin concentration during the study (pmol/L)
Glucose concentration | Through study completion, within 2 years
  Glucose concentration during the study (mmol/L)
Cortisol concentration | Through study completion, within 2 years
  Cortisol concentration during the study (ng/L)

OTHER OUTCOMES:
Weight | Through study completion, within 2 years
  Participant weight (kg)
Height | Through study completion, within 2 years
  Participant height (cm)
BMI | Through study completion, within 2 years
  BMI is measured as weight (kg)/height squared (m2) (kg/m2 squared)
HbA1c | Through study completion, within 2 years
  Hemoglobin A1c (mmol/mol of Hemoglobulin )
Age | at Screening visit
  Age (y)
Systolic blood pressure | Through study completion, within 2 years
  Systolic blood pressure (mmHg)
Diastolic blood pressure | Through study completion, within 2 years
  Diastolic blood pressure (mmHg)
Heart beat (BP) | Through study completion, within 2 years
  Heart beat (BP) bpm

CONTACTS AND LOCATIONS:
Locations (1):
- David L. Russell-Jones, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available following the statistical analysis 2/01/2025
Access Criteria: Once the data is avalible

REFERENCES:
- [Result] Fan KS, Shojaee-Moradie F, Manoli A, Baumann PM, Koehler G, Edwards V, Lee V, Mathieu C, Mader JK, Russell-Jones D; EASA Diabetes Consortium. The Feasibility of an Experimental Hypobaric Simulation to Evaluate the Safety of Closed-Loop Insulin Delivery Systems in Flight-Related Atmospheric Pressure Changes. Diabetes Technol Ther. 2025 Feb;27(2):128-133. doi: 10.1089/dia.2024.0380. Epub 2024 Oct 24. PMID 39446977
- [Result] Fan KS, Manoli A, Shojaee-Moradie F, Hutchison E, Strollo F, Koehler G, Mader JK, Russell-Jones D; EASA Diabetes Consortium. The practical operation and consequences of glucose measurement by pilots with diabetes. Diabet Med. 2025 Mar;42(3):e15472. doi: 10.1111/dme.15472. Epub 2024 Nov 9. PMID 39521725
- [Result] Garden GL, Fan KS, Paterson M, Shojaee-Moradie F, Borg Inguanez M, Manoli A, Edwards V, Lee V, Frier BM, Hutchison EJ, Maher D, Mathieu C, Mitchell SJ, Heller SR, Roberts GA, Shaw KM, Koehler G, Mader JK, King BR, Russell-Jones DL; EASA Diabetes Consortium. Effects of atmospheric pressure change during flight on insulin pump delivery and glycaemic control of pilots with insulin-treated diabetes: an in vitro simulation and a retrospective observational real-world study. Diabetologia. 2025 Jan;68(1):52-68. doi: 10.1007/s00125-024-06295-1. Epub 2024 Nov 4. PMID 39496965